CLINICAL TRIAL: NCT06650579
Title: Randomized Controlled Trial of Leuprolide Plus Abiraterone Acetate (AA) Versus Relugolix Plus AA for Advanced Prostate Cancer: The REVELUTION-2 Trial
Brief Title: REVELUTION-2: Relugolix+Abiraterone Acetate (AA) Versus Leuprolide+AA Cardiac Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry); Sumitomo Pharma America, Inc. (Industry); National Comprehensive Cancer Network (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sagar Patel, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00007557; P30CA138292 (NIH); NCI-2024-07761 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007557 (Other: Emory University Hospital); RAD6197-24 (Other: Emory University Hospital)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Prostate Carcinoma; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
Keywords: node-positive prostate cancer; advanced prostate cancer; very-high-risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; bicalutamide; Specimen Handling; Leuprolide; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; relugolix

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All principal investigators and co-investigators will be blinded to randomization block. All cardiac computed tomography images will be analyzed by a blinded level 3 boarded cardiac imaging expert.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (leuprolide plus abiraterone acetate/prednisone) (Experimental): Patients receive leuprolide IM or SC injections every 3 to 6 months plus oral abiraterone acetate (AA) with prednisone daily for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy.
  Interventions: Drug: Abiraterone Acetate; Drug: Bicalutamide; Procedure: Biospecimen Collection; Procedure: Computed Tomography Angiography; Drug: Leuprolide; Drug: Prednisone; Radiation: Radiation Therapy
- Arm II (relugolix + abiraterone acetate/prednisone) (Experimental): Patients receive oral relugolix daily plus oral abiraterone acetate (AA) with prednisone daily for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy.
  Interventions: Drug: Abiraterone Acetate; Procedure: Biospecimen Collection; Procedure: Computed Tomography Angiography; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Relugolix

INTERVENTIONS:
Drug: Abiraterone Acetate — Given abiraterone acetate
  Other Names: BR9004; BR9004-1; CB 7630; CB-7630; CB7630; JNJ-212082; Yonsa; Zytiga
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cassotide; Cosudex; ICI 176,334; ICI 176334; Utamide
  Arms: Arm I (leuprolide plus abiraterone acetate/prednisone)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography Angiography — Undergo CCTA
  Other Names: CT ANGIOGRAPHY; CT Scan Angiography; CTA
Drug: Leuprolide — Given IM or SC
  Other Names: Leuprorelin
  Arms: Arm I (leuprolide plus abiraterone acetate/prednisone)
Drug: Prednisone — Given prednisone
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Undergo standard of care radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Relugolix — Given PO
  Other Names: N-(4-(1-((2,6-Difluorophenyl)methyl)-5-((dimethylamino)methyl)-1,2,3,4-tetrahydro-3-(6-methoxy-3-pyridazinyl)-2,4-dioxothieno(2,3-d)pyrimidin-6-yl)phenyl)-N'-methoxyurea; Orgovyx; Relumina; TAK 385; TAK-385; TAK385
  Arms: Arm II (relugolix + abiraterone acetate/prednisone)

SUMMARY:
This phase III/IV trial compares the impact of leuprolide and abiraterone acetate (AA) versus relugolix and AA on the heart in hormone-naive patients with advanced prostate cancer receiving pelvic radiation therapy. Leuprolide is in a class of medications called gonadotropin-releasing hormone agonists (GNRHa). It prevents the body from making luteinizing hormone-releasing hormone (LHRH) and luteinizing hormone (LH). This causes the testicles to stop making testosterone (a male hormone) in men and may stop the growth of prostate tumor cells that need testosterone to grow. Abiraterone acetate, an androgen biosynthesis inhibitor, works by decreasing the amount of certain hormones in the body. Relugolix, a GNRH antagonist, works by decreasing the amount of testosterone produced by the body. This may slow or stop the spread of prostate tumor cells that need testosterone to grow. The use of hormone therapy with radiation therapy has been shown to improve survival, however, studies have suggested that the addition of hormone therapy may worsen heart (cardiac) disease and high blood pressure. In fact, studies have shown that the most common cause of death in prostate cancer patients is due to heart disease or heart attacks. Computed tomography (CT) scans create a series of detailed pictures of areas inside the body; the pictures are created by a computer linked to an x-ray machine. In this study, sophisticated cardiac CT images are used to take pictures of patients' heart and coronary arteries to help assess damage to the heart. Using cardiac CT and blood tests, this trial may help doctors determine which patients are at risk of cardiac disease when treated with combination hormone therapy, as well as the differential risk of leuprolide versus relugolix in combination with abiraterone acetate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Measure cardiovascular outcomes between combination gonadotropin releasing hormone agonist (GNRHa, i.e. leuprolide) plus abiraterone acetate (AA) versus gonadotropin releasing hormone antagonist (GNRH-antagonist, i.e. relugolix) plus AA in men with advanced prostate cancer receiving definitive radiation therapy.

SECONDARY OBJECTIVES:

I. Identify genomic alterations that predispose an individual to enhanced cardiovascular (CV) toxicity following hormone therapy with leuprolide or relugolix in combination with abiraterone acetate.

II. Evaluate serum testosterone kinetics during and after treatment with combination leuprolide+AA versus relugolix+AA.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive leuprolide intramuscularly (IM) or subcutaneously (SC) injection every 3 to 6 months plus oral AA with prednisone daily for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy. Patients may also receive bicalutamide orally (PO) once daily (QD) on days 21-30 with first injection of leuprolide at the discretion of the treating provider. All patients undergo pre-treatment and 12-month coronary computed tomography angiography (CCTA) and blood sample collection.

ARM II: Patients receive oral relugolix PO daily plus oral AA with prednisone daily for up to 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo standard of care radiation therapy. All patients undergo pre-treatment and 12-month CCTA and blood sample collection.

After completion of study treatment, patients are followed up at 30 and 60 days for serum testosterone measurement.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years old
* Non-metastatic prostate cancer
* Non-metastatic, biochemically recurrent prostate cancer
* Plan to undergo curative-intent pelvic radiation therapy (photons or protons) with or without brachytherapy
* Plan to undergo up to 24 months of combination androgen deprivation therapy (ADT) plus AA and prednisone

Exclusion Criteria:

* Metastatic prostate cancer requiring indefinitive ADT or chemotherapy
* Prior exposure to androgen deprivation therapy
* Prior exposure to chemotherapy, immunotherapy, or radiation therapy
* History of cardiac bypass surgery or percutaneous coronary intervention
* History of cardiac pacemaker or defibrillator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of ambulatory systolic blood pressure (BP) > 140 or diastolic > 90 (measurement on 2 separate days) | At baseline and up to 12 months
  The change will be estimated and tested using paired tests (Wilcoxon signed rank test or McNemar test). The difference at each interval for the two groups will be tested using Fisher's exact test for binary endpoints or Wilcoxon rank-sum test for continuous. Data transformation to fit statistical assumptions will be done as needed. Multivariable models that control for potential confounders will be implemented using general linear and logistic regression.
Need for new or escalated anti-hypertensive medication | At baseline and up to 12 months
  The change will be estimated and tested using paired tests (Wilcoxon signed rank test or McNemar test). The difference at each interval for the two groups will be tested using Fisher's exact test for binary endpoints or Wilcoxon rank-sum test for continuous. Data transformation to fit statistical assumptions will be done as needed. Multivariable models that control for potential confounders will be implemented using general linear and logistic regression.
Incidence of moderate-to-severe atherosclerosis of major coronary vessels | From month 0 to month 12
  Defined as > 50% luminal stenosis per the Society of Cardiac Computed Tomography. Change will be tested using paired tests (Wilcoxon signed rank test or McNemar test). Luminal stenosis will be measured on a per-vessel basis. Proportion of patients achieving > 50% luminal stenosis of a major coronary vessel between each arm will be compared using Fisher's exact test. The percent change of maximal stenosis between the two arms will be tested using Wilcoxon signed rank test.

SECONDARY OUTCOMES:
Total plaque volume | From month 0 to month 12
  Total plaque volume (per-patient and per-vessel basis, respectively) will be measured. Adjusted mean difference will be calculated from baseline to month 12 between arms. Multivariable adjustment will be utilized that control age and statin using logistic regression.
Pre-existing genomic alterations promoting inflammatory immunity and associated with cardiovascular disease | At baseline
  Pre-treatment samples will be subjected to whole exome sequencing to determine alterations to the protein-coding regions of the genome, specifically those associated with clonal hematopoiesis of indeterminate potential (CHIP). The association of CHIP mutations with development of cardiovascular toxicity following therapy will be measured.
Castration rate | At study days 7, 30 and 90
  The cumulative probability of testosterone suppression to ≤ 50 ng/dL will be summarized using the Kaplan-Meier method. Confidence intervals will be calculated using the exponential Greenwood formulation via log-log transformation of the survival function
Sustained castration | At months 6 and 12
  The probability of testosterone suppression ≤ 50 ng/mL will be summarized using Kaplan-Meier. Confidence intervals will be calculated using the exponential Greenwood formulation via log-log transformation of the survival function
Testosterone recovery | At day 30 and/or day 90 following completion of androgen deprivation therapy
  The probability of testosterone recovery > 50 ng/mL and 200 ng/mL will be summarized using the Kaplan-Meier method. Confidence intervals will be calculated using the exponential Greenwood formulation via log-log transformation of the survival function

CONTACTS AND LOCATIONS:
Overall Officials: Sagar A Patel, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Winship at Emory Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia